CLINICAL TRIAL: NCT02065180
Title: The Effect of a Red Rice and Olive Extract Nutrition Supplement on Cholesterol
Brief Title: The Effect of a Red Rice and Olive Extract Nutrition Supplement on Cholesterol Levels in Patients With Metabolic Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Veronique Verhoeven, Professor, Universiteit Antwerpen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: verhoevenhermans
Record Dates: First submitted 2014-02-13; First posted 2014-02-17 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Hypercholesterolaemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- commercially available nutrition supplement (Experimental): this group receives a commercially available nutritional supplement for a period of 2 months
  Interventions: Dietary Supplement: commercially available nutrition supplement
- control group (Placebo Comparator): this group receives a placebo for a period of 2 months
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: commercially available nutrition supplement — the food supplement contains red rice yeast and olive extract
  Arms: commercially available nutrition supplement
Dietary Supplement: placebo
  Arms: control group

SUMMARY:
This randomised controlled trial studies the effect of a commercially available nutritional supplement on cholesterol levels in people with metabolic syndrome and elevated cholesterol levels.

ELIGIBILITY:
Inclusion Criteria:

* metabolic syndrome according to ATPIII criteria 3 of the following:

  * waist circumference >88cm (in females) or >102cm (in males)
  * triglycerides >150mg/dl
  * HDL <40 (50)mg/dl in males (females)
  * blood pressure>130/85 or treatment for AHT
  * glucose >110mg/dl

Exclusion Criteria:

* pregnancy
* treatment with cholesterol lowering drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
LDL level | 2 months
total cholesterol level | 2 months
triglyceride level | 2 months
HDL level | 2 months

SECONDARY OUTCOMES:
OxLDL | 2 months
BMI | 2 months
malondialdehyde (MDA) | 2 months
8-OH-deoxyguanosine (8-OHdG) | 2 months
side effects | 2 months
waist circumference | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Antwerp, Antwerp, Belgie, Belgium

REFERENCES:
- [Derived] Hermans N, Van der Auwera A, Breynaert A, Verlaet A, De Bruyne T, Van Gaal L, Pieters L, Verhoeven V. A red yeast rice-olive extract supplement reduces biomarkers of oxidative stress, OxLDL and Lp-PLA2, in subjects with metabolic syndrome: a randomised, double-blind, placebo-controlled trial. Trials. 2017 Jul 3;18(1):302. doi: 10.1186/s13063-017-2058-5. PMID 28673363
- [Derived] Verhoeven V, Van der Auwera A, Van Gaal L, Remmen R, Apers S, Stalpaert M, Wens J, Hermans N. Can red yeast rice and olive extract improve lipid profile and cardiovascular risk in metabolic syndrome?: A double blind, placebo controlled randomized trial. BMC Complement Altern Med. 2015 Mar 10;15:52. doi: 10.1186/s12906-015-0576-9. PMID 25879228